CLINICAL TRIAL: NCT03889275
Title: An Open-label Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of MEDI5395 in Combination With Durvalumab in Subjects With Select Advanced Solid Tumors.
Brief Title: A Study of MEDI5395 in Combination With Durvalumab in Participants With Select Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6450C00001
Record Dates: First submitted 2019-03-08; First posted 2019-03-26 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumors
Keywords: solid tumors; immunotherapy; oncolytic virus; NDV-GMCSF
MeSH Terms: interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1A: MEDI5395 Dose Level 1 + Sequential Durvalumab (Experimental): Participants will receive IV infusions of MEDI5395 Dose Level 1 on Days 1, 4, 8, 10, 12, and 15 followed by durvalumab every 4 weeks (Q4W) starting from 14 days after the last dose of MEDI5395 for maximum of 2 years or until disease progression, clinical deterioration, withdrawal of consent, or unacceptable toxicity; whichever occurs first.
  Interventions: Biological: MEDI5395; Biological: Durvalumab
- Cohort 2A: MEDI5395 Dose Level 2 + Sequential Durvalumab (Experimental): Participants will receive IV infusions of MEDI5395 Dose Level 2 on Days 1, 4, 8, 10, 12, and 15 followed by durvalumab Q4W starting from 14 days after the last dose of MEDI5395 for maximum of 2 years or until disease progression, clinical deterioration, withdrawal of consent, or unacceptable toxicity; whichever occurs first.
  Interventions: Biological: MEDI5395; Biological: Durvalumab
- Cohort 3A: MEDI5395 Dose Level 3 + Sequential Durvalumab (Experimental): Participants will receive IV infusions of MEDI5395 Dose Level 3 on Days 1, 4, 8, 10, 12, and 15 followed by durvalumab Q4W starting from 14 days after the last dose of MEDI5395 for maximum of 2 years or until disease progression, clinical deterioration, withdrawal of consent, or unacceptable toxicity; whichever occurs first.
  Interventions: Biological: MEDI5395; Biological: Durvalumab
- Cohort 3A Backfill: MEDI5395 Dose Level 3 + Sequential Durvalumab (Experimental): Participants will receive IV infusions of MEDI5395 Dose Level 2 on Day 1 and Dose Level 3 on Days 4, 8, 10, 12, and 15 followed by durvalumab Q4W starting from 14 days after the last dose of MEDI5395 for maximum of 2 years or until disease progression, clinical deterioration, withdrawal of consent, or unacceptable toxicity; whichever occurs first.
  Interventions: Biological: MEDI5395; Biological: Durvalumab
- Cohort 4A: MEDI5395 Dose Level 4 + Sequential Durvalumab (Experimental): Participants will receive IV infusions of MEDI5395 Dose Level 2 on Day 1 and Dose Level 4 on Days 4, 8, 10, 12, and 15 followed by durvalumab Q4W starting from 14 days after the last dose of MEDI5395 for maximum of 2 years or until disease progression, clinical deterioration, withdrawal of consent, or unacceptable toxicity; whichever occurs first.
  Interventions: Biological: MEDI5395; Biological: Durvalumab
- Cohort 1B: MEDI5395 Dose Level 1 + Concurrent Durvalumab (Experimental): Participants will receive IV infusions of MEDI5395 Dose Level 1 on Days 1, 4, 8, 10, 12, and 15 and durvalumab Q4W, starting from the same day as third dose of MEDI5395, for maximum of 2 years or until disease progression, clinical deterioration, withdrawal of consent, or unacceptable toxicity; whichever occurs first.
  Interventions: Biological: MEDI5395; Biological: Durvalumab
- Cohort 2B: MEDI5395 Dose Level 2 + Concurrent Durvalumab (Experimental): Participants will receive IV infusions of MEDI5395 Dose Level 2 on Days 1, 4, 8, 10, 12, and 15 and durvalumab Q4W, starting from the same day as third dose of MEDI5395, for maximum of 2 years or until disease progression, clinical deterioration, withdrawal of consent, or unacceptable toxicity; whichever occurs first.
  Interventions: Biological: MEDI5395; Biological: Durvalumab
- Cohort 3B: MEDI5395 Dose Level 3 + Concurrent Durvalumab (Experimental): Participants will receive IV infusions of MEDI5395 Dose Level 3 on Days 1, 4, 8, 10, 12, and 15 and durvalumab Q4W, starting from the same day as third dose of MEDI5395, for maximum of 2 years or until disease progression, clinical deterioration, withdrawal of consent, or unacceptable toxicity; whichever occurs first.
  Interventions: Biological: MEDI5395; Biological: Durvalumab

INTERVENTIONS:
Biological: MEDI5395 — Participants will receive multiple dose levels of MEDI5395 over several days as stated in arm description.
Biological: Durvalumab — Participants will receive IV infusion of durvalumab as stated in arm description.
  Other Names: Imfinzi

SUMMARY:
The reason for the study is to find out if MEDI5395 and durvalumab will work and be safe for the treatment of solid tumors.

DETAILED DESCRIPTION:
This is an Phase 1, first-in-human, open-label, dose-escalation, and dose-expansion study to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics and preliminary efficacy of MEDI5395 in combination with durvalumab in participants with selected advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria

* The participant must consent to take precautionary measures to prevent Newcastle Disease Virus (NDV) transmission to humans and birds
* Participants must have histologic documentation of advanced solid tumor and received and have progressed, are refractory, or are intolerant to standard therapy for the specific tumor type. All participants are required to have had at least one prior line of treatment in the recurrent or metastatic setting
* Participants must have at least 1 measurable lesion and an additional non-lymph node non-target lesion that can be biopsied at acceptable risk as judged by the investigator. (Note: if a non-target lesion is not available or cannot be biopsied, a RECIST target, non-lymph node lesion, lesion >= 2 cm in longest diameter may be used for non-excisional biopsy
* All participants must consent to provide tumor tissue for correlative studies
* The ECOG performance status of 0 to 1
* Adequate organ function
* Use of highly effective contraception (females) or male condom plus spermicide (males)

Exclusion Criteria

* Rapidly progressing disease defined as a participant that cannot tolerate a break of at least 8 weeks from systemic anticancer therapy.
* Primary central nervous system (CNS) disease is excluded
* Participants who have received prior check point inhibitor immunotherapy within 28 days and/or oncolytic virus therapy within 90 days prior to the first dose of MEDI5395
* Unresolved toxicities from prior anticancer therapy that led to permanent discontinuation of prior immunotherapy or that required immunosuppression other than corticosteroids
* History of severe allergic reactions to any of the study drug components
* Infectious disease exclusions including tuberculosis, Human immunodeficiency virus (HIV), hepatitis A, B or C, active bacterial, fungal or viral infections plus receipt of live attenuated vaccine prior to first dose of MEDI5395. (NOTE: Participants with evidence of fully recovered past hepatitis B infection who developed immunity OR hepatitis B/C with undetectable virus load and are on medications may be permitted).
* Positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) diagnostic test at screening
* Any conditions requiring use of any systemic immunosuppressant including systemic corticosteroids, methotrexate, azathioprine, tumor necrosis factor (TNF) inhibitor, and/or interleukin 6 (IL-6) blockers
* Active autoimmune disease or chronic inflammatory condition (Exceptions include vitiligo, alopecia, hypothyroidism on stable treatment, diverticulosis, controlled celiac disease, and chronic skin conditions not requiring systemic therapy)
* Active acquired immune-deficiency states
* Participants who are regularly exposed to poultry or birds
* Current active hepatitis or biliary disease (except for Gilbert's syndrome, asymptomatic gallstones, or stable chronic liver disease)
* Clinically significant pulmonary disease and cardiac disease
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of participant safety or study results.

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) | From first dose of MEDI5395 through 14.4 months (corresponding to maximum observed duration)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Number of Participants with Dose-limiting Toxicities (DLT) | Day 1 to Day 28 of first dose of MEDI5395
  A DLT is defined as any toxicity not clearly and directly related to the primary disease or to another etiology and included: any Grade 3 or higher toxicity that occurs during the DLT evaluation period, aspartate aminotransferase or alanine aminotransferase >= 3 × upper limit of normal (ULN) together with total bilirubin >= 2 × ULN, where no other reason other than the study drugs, can be found to explain the combination of increases, Grade ≥ 2 myocarditis, Grade 2 non infectious pneumonitis that does not resolve to Grade ≤ 1 within 7 days of the initiation of maximal supportive care, any Grade >= 2 MEDI5395 related toxicity that prevents administration of more than 1 dose of MEDI5395 within the 18-day dosing period, in sequential dosing cohorts, any Grade >= 2 MEDI5395 related toxicity that prevents administration of the first dose of durvalumab, and any AE that, after consultation with the Sponsor and investigators, is deemed a DLT.
Number of Participants with TEAEs Resulting in Permanent Discontinuation of MEDI5395 | From first dose of MEDI5395 through 14.4 months (corresponding to maximum observed duration)
  Number of participants with TEAEs resulting in permanent discontinuation of MEDI5395 are reported.
Number of Participants with TEAEs Resulting in Permanent Discontinuation of Durvalumab | From first dose of durvalumab through 14.4 months (corresponding to maximum observed duration)
  Number of participants with TEAEs resulting in permanent discontinuation of durvalumab are reported.
Number of Participants With Abnormal Vital Signs Reported as TEAEs | From first dose of MEDI5395 through 14.4 months (corresponding to maximum observed duration)
  Number of participants with abnormal vital signs (blood pressure, pulse rate, respiration rate, oxygen saturation, and body temperature) reported as TEAEs are reported.
Number of Participants With Abnormal Laboratory Parameters Reported as TEAEs | From first dose of MEDI5395 through 14.4 months (corresponding to maximum observed duration)
  Laboratory assessment included hematology, clinical chemistry, coagulation, cardiac parameters, and urinalysis. Participants with abnormal laboratory parameters reported as TEAEs are reported.
Number of Participants With Abnormal Electrocardiogram (ECG) Parameters Reported as TEAEs | From first dose of MEDI5395 through 14.4 months (corresponding to maximum observed duration)
  Number of participants with abnormal ECG parameters reported as TEAEs are reported.
Change From Baseline in Left Ventricular Ejection Fraction (LVEF) | From first dose of MEDI5395 through 14.4 months (corresponding to maximum observed duration)
  Change from baseline in LVEF values are reported.
Maximum Reduction From Baseline in Global Longitudinal Strain (GLS) Values | From first dose of MEDI5395 through 14.4 months (corresponding to maximum observed duration)
  Maximum reduction from baseline in GLS values are reported. The GLS < 16% is abnormal, GLS > 18% is normal, and GLS 16% to 18% is borderline.
Number of Participants With at Least 1-Grade Shift From Baseline to Worst Post-baseline in Eastern Co-operative Oncology Group Performance Status (ECOG-PS) Score | From first dose of MEDI5395 through 14.4 months (corresponding to maximum observed duration)
  ECOG performance status is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. The scores are: 0 = Fully Active, able to carry out all pre-disease performance without restrictions; 1 = Restricted activity but ambulatory and able to carry out light work or work of a sedentary nature; 2 = Ambulatory and capable of self-care but unable to carry out work activities; 3 = Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4 = Completely Disabled, unable to carry out any self-care and totally confined to bed or chair; 5 = Dead.

SECONDARY OUTCOMES:
Percentage of Participants with Objective Response per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | Baseline (Day -28 to Day -1) through 24.5 months (corresponding to maximum observed duration)
  The OR is defined as confirmed complete response (CR) or confirmed partial response (PR) based on RECIST v1.1 guidelines. The CR is defined as disappearance of all target and non-target lesions and normalization of tumor marker level and all lymph nodes (target and non-target) must be non-pathological in size (< 10 mm in short axis). The PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. A confirmed CR or PR is defined as 2 CRs or 2 PRs that were separated by at least 4 weeks with no evidence of progression in-between.
Percentage of Participants with Disease Control (DC) per RECIST v1.1 | Baseline (Day -28 to Day -1) through 24.5 months (corresponding to maximum observed duration)
  The DC is confirmed CR, PR, or stable disease (SD) per RECIST v1.1 guidelines. The CR is defined as disappearance of all target and non-target lesions (TLs and NTLs), normalization of tumor marker level, all lymph nodes (target and non-target) must be non-pathological in size (<10 mm in short axis), and no new lesions. The PR is defined as at least a 30% decrease in sum of diameters (SoD) of TLs, taking as reference the baseline SoD and no new NTL. A confirmed CR or PR is defined as 2 CRs or 2 PRs that were separated by at least 4 weeks with no evidence of progression in-between. The SD is defined as neither sufficient shrinkage of TLs to qualify for PR nor sufficient increase of TLs to qualify for progressive disease (PD), taking as reference the smallest SoD while on study and no new lesions. The PD is defined as at least a 20% increase in SoD of TLs, taking as reference the smallest sum on study and an absolute increase of at least 5 mm of SoD, or the appearance of new lesions.
Duration of Response (DoR) per RECIST v1.1 | Baseline (Day -28 to Day -1) through 24.5 months (corresponding to maximum observed duration)
  DoR: Time from first documentation of OR to first documented PD or death due to any cause, whichever occurred first. OR: Confirmed CR or confirmed PR based on RECIST v1.1 guidelines. CR: Disappearance of all target and non-target lesions, normalization of tumor marker level, all lymph nodes (target and non-target) must be non-pathological in size (< 10 mm in short axis), and no new lesions. PR: At least a 30% decrease in the SoD of target lesions, taking as reference the baseline sum diameters and no new lesions. A confirmed CR or PR is defined as 2 CRs or 2 PRs that were separated by at least 4 weeks with no evidence of progression in-between. PD: At least a 20% increase in SoD of target lesion, taking as reference the smallest sum on study and an absolute increase of at least 5 mm of sum of diameters, or the appearance of new lesions. The DOR is estimated using the Kaplan-Meier method.
Time to Response (TTR) per RECIST v1.1 | Baseline (Day -28 to Day -1) through 24.5 months (corresponding to maximum observed duration)
  The TTR is defined as the time from the start of treatment with any study drug until the first documentation of a subsequently confirmed OR. The OR is defined as confirmed CR or confirmed PR based on RECIST v1.1 guidelines. The CR is defined as disappearance of all target and non-target lesions, normalization of tumor marker level, all lymph nodes (target and non-target) must be non-pathological in size (< 10 mm in short axis), and no new lesions. The PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters and no new lesions. A confirmed CR or PR is defined as 2 CRs or 2 PRs that were separated by at least 4 weeks with no evidence of progression in-between. The TTR is assessed using the Kaplan-Meier method.
Progression-Free Survival (PFS) per RECIST v1.1 | Baseline (Day -28 to Day -1) through 24.5 months (corresponding to maximum observed duration)
  The PFS is defined as the time from the start of treatment with any study drug until the first documentation of disease progression or death due to any cause, whichever occurred first. Disease progression is defined as at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study and an absolute increase of at least 5 mm of sum of diameters, or the appearance of one or more new lesions. The PFS is estimated using the Kaplan-Meier method.
Overall Survival (OS) | Baseline (Day -28 to Day -1) through 24.5 months (corresponding to maximum observed duration)
  The OS is defined as the time from the start of treatment with study drug until death due to any cause. The OS is estimated using the Kaplan-Meier method.
Viral Genome Concentration of MEDI5395 in Whole Blood | Predose and end of infusion; on dose 1,2,3,4,5,6, 1 day(D) post Dose 1 and 6, 7 D post Dose 6 of MEDI5395/Cycle(C)1D15, C2D1, C3D1,C4D1, and C5D1 pre dose of durvalumab in both sequential and concurrent dosing; C1D1, C1D8, and C1D15 in sequential dosing
  Viral genome concentration of MEDI5395 in whole blood is reported.
Number of Participants With Positive Neutralizing Antibodies (nAbs) to MEDI5395 | Day (D) of MEDI5395 (MEDI) Dose 1, 4, 6, D1 C1 and C2 of durvalumab in sequential dosing; on day of MEDI Dose 1, 4, 6; C1D15, C2D1 C3D1, C4D1 of durvalumab dose in concurrent dosing; within 28 days of last dose (LD) and 90 days post LD (14.4 months)
  Number of participants with positive nAbs to MEDI5395 are reported. Persistent positive is defined as positive at >=2 post-baseline assessments (with >=16 weeks between first and last positive assessment) or positive at last post-baseline assessment. Transient positive is defined as negative at the last post-baseline assessment and positive at only 1 post-baseline assessment or at >= 2 post-baseline assessments (with < 16 weeks between the first and last positive assessment).
Tumoral Cluster of Differentiation 8 Positive (CD8+) Cell Density in Tumor Tissue | Baseline (Pre-treatment) and on the Day of Dose 4 of MEDI5395 (Post-treatment)
  The CD8+ cells were assessed by validated immunohistochemical (IHC) assays using tumor tissue from an archival or newly obtained biopsy. The results of CD8+ cell density was reported as number of CD8+ positive cells per mm^2.
Percentage of Programmed Cell Death Ligand 1 (PD-L1) Positivity in Tumor Cells | Baseline (Pre-treatment) and on the Day of Dose 4 of MEDI5395 (Post-treatment)
  The PD-L1 expression was assessed by validated IHC assays using tumor tissue from an archival or newly obtained biopsy. Tumor cells were analyzed for PD-L1 expression to determine the tumor cells positivity for PD-L1.
Percentage of PD-L1 Positvity in Whole Biopsy Sample | Baseline (Pre-treatment) and on the Day of Dose 4 of MEDI5395 (Post-treatment)
  The PD-L1 expression was assessed by validated IHC assays using tumor tissue from an archival or newly obtained biopsy. The whole biopsy sample (without differentiation between tumor or stromal/immune compartments) was analyzed for PD-L1 expression to determine total tissue positivity (TIP) for PD-L1.

CONTACTS AND LOCATIONS:
Overall Officials: Medimmune LLC, Study Director — MedImmune LLC
Locations (10):
- United States (8):
  - Research Site, Phoenix, Arizona
  - Research Site, La Jolla, California
  - Research Site, Rochester, Minnesota
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Providence, Rhode Island
- United Kingdom (2):
  - Research Site, Leeds
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Davar D, Carneiro BA, Dy GK, Sheth S, Borad MJ, Harrington KJ, Patel SP, Galanis E, Samson A, Agrawal S, Chen Z, Fan C, Gong M, Burton J, Tu E, Durham N, Laubscher K, Arnaldez F, Zamarin D. Phase I study of a recombinant attenuated oncolytic virus, MEDI5395 (NDV-GM-CSF), administered systemically in combination with durvalumab in patients with advanced solid tumors. J Immunother Cancer. 2024 Nov 17;12(11):e009336. doi: 10.1136/jitc-2024-009336. PMID 39551600
- See also: CSR Synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6450C00001&attachmentIdentifier=8c5b1e69-7c75-4dd2-bc86-5f8d988c2fa1&fileName=D6450C00001-study-synopsis_final-Redacted.pdf&versionIdentifier=